CLINICAL TRIAL: NCT04986371
Title: An Observational, Non-interventional Study of Niraparib Maintenance Treatment in Patients With Ovarian Cancer After Frontline Platinum-based Chemotherapy
Brief Title: Real-world Study of Niraparib Maintenance Treatment in Patients With Newly Diagnosed Ovarian Cancer
Acronym: RENI-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ling-Ying Wu (Unknown)
Responsible Party: Sponsor-Investigator, Ling-Ying Wu, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: 21/251-2922
Record Dates: First submitted 2021-07-16; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — niraparib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue, peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Niraparib — Usage following drug insert is recommended
  Other Names: Zejula

SUMMARY:
This is an open-label, single-arm, multi-center、non-interventional real-world study, which evaluate treatment pattern, safety and efficacy of Niraparib as first-line maintenance treatment for Chinese patient with newly diagnosed ovarian cancer , fallopian tube cancer, and primary peritoneal cancer in real world clinical practice.

DETAILED DESCRIPTION:
In this study, 300 patients will be enrolled. Eligible patients will be those with histologically confirmed epithelial ovarian cancer, carcinoma of fallopian tube or primary peritoneal carcinoma. Patients must have received one line of platinum-based chemotherapy, and be in clinically complete or partial response following the platinum-based chemotherapy prior to enrollment in the study. Patients will be treated with Niraparib according to the physician's judgement till disease progression, discontinuation for other reasons or death. The primary endpoint is treatment pattern of Niraparib as first-line maintenance treatment for ovarian cancer patients. The second endpoints include AE, PFS and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Histologically confirmed epithelial ovarian cancer, carcinoma of fallopian tube or primary peritoneal carcinoma
* Having received one line of platinum-based chemotherapy, and clinically CR or PR to this line of chemotherapy
* Understand the protocol, and Written informed consent before any study-related procedure

Exclusion Criteria:

* Participating in other clinical trials at the same time
* Having sever or uncontrolled diseases that will influence the study, according to the judgement of investigators
* Having other malignant tumors (other than breast cancer with BRCA mutation)
* Pregnancy or breast feeding, or planning a pregnancy during the study
* Unable to visit on time
* Patients who are allergic to the study drug or drug components

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-10 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Starting dose of Niraparib | up to 3 years
  Record the starting dose of Niraparib in real clinical practice
Percentage of patients who have taken dose adjustment and the reason of dose adjustment | up to 3 years
  Record the percentage of patients who have taken dose adjustment and the reason of dose adjustment
Percentage of patients who have taken dose discontinuation and the reason of dose discontinuation | up to 3 years
  Record the percentage of patients who have taken dose discontinuation and the reason of dose discontinuation
Concomitant treatments which patients take along with Niraparib | up to 3 years
  Record the concomitant treatments (drugs, or other tumor treatments) which patients take along with Niraparib

SECONDARY OUTCOMES:
Incidence of all AEs | up to 3 years
  Incidence of all AEs based upon CTCAE version 5.0 during subjects receiving the study treatment.
Progression-free survival (PFS) | up to 3 years
  Progression-free survival is defined as the time from the last day of previous chemotherapy to first documentation of tumor progression, or to death due to any cause in the absence of previous documentation of objective tumor progression.
Time to First Subsequent Therapy (TFST) | up to 3 years
  The TFST was defined as the time from the last day of previous chemotherapy to the start date of the first subsequent anti-cancer therapy or death.
Chemotherapy-Free Interval (CFI) | up to 3 years
  CFI was defined as the time to the initiation of the next anti-cancer therapy after maintenance treatment.
Overall Survival (OS) | up to 3 years
  Overall survival is defined as the date of the last day of previous chemotherapy to the date of death by any cause.
Change From Baseline in EQ-5D-5L | up to 3 years
  EQ-5D-5L is a well-validated, general preference-based, health-related QoL instrument. The EQ-5D-5L encompasses 5 domains, asking patients to rate their perceived health state today on the following dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each domain has 5 possible levels: "no problems" (Level 1), "slight problems" (Level 2), "moderate problems" (Level 3), "severe problems" (Level 4), and "extreme problems" (Level 5). Each domain is assigned a level, and levels are combined to create a 5-digit number describing the patient's health state. For each patient, an index value is determined from a published country-specific value set. This index value or utility score ranges from 0 to 1.00 (with 1.0 representing perfect health) and is used in the calculation of quality-adjusted life years (QALYs) that are used to inform economic valuations of health interventions. A positive change from baseline indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Lingying Wu, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No